CLINICAL TRIAL: NCT01894568
Title: A Phase 3, Open Label, Randomized, Parallel, 26 Week Treatment Study Comparing LY2605541 With Insulin Glargine as Basal Insulin Treatment in Combination With Oral Anti Hyperglycemia Medications in Asian Insulin Naïve Patients With Type 2 Diabetes Mellitus
Brief Title: A Study Comparing Insulin Peglispro With Insulin Glargine as Basal Insulin Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13422; I2R-JE-BIAQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — basal insulin peglispro; LY2605541; Insulin Glargine; Sulfonylurea Compounds; meglitinide; Dipeptidyl Peptidase 4; Biguanides; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Peglispro (Experimental): Insulin Peglispro administered subcutaneously (SC) once daily for 26 weeks in combination with Oral Antihyperglycemic Medications (OAMs).
  Interventions: Drug: Insulin Peglispro; Drug: Oral Antihyperglycemic Medications (OAMs)
- Insulin Glargine (Active Comparator): Insulin Glargine administered SC once daily for 26 weeks in combination with OAMs.
  Interventions: Drug: Insulin Glargine; Drug: Oral Antihyperglycemic Medications (OAMs)

INTERVENTIONS:
Drug: Insulin Peglispro — Administered SC using a prefilled pen.
  Other Names: LY2605541
  Arms: Insulin Peglispro
Drug: Insulin Glargine — Administered SC using a prefilled pen
  Arms: Insulin Glargine
Drug: Oral Antihyperglycemic Medications (OAMs) — Administered orally
  Other Names: Sulfonylureas; Meglitinides; Dipeptidyl Peptidase-4 (DPP-IV) Inhibitors; Biguanides; α-Glucosidase Inhibitors; Pioglitazone

SUMMARY:
The purpose of this study is to compare insulin peglispro (LY2605541) to insulin glargine in Asian insulin naïve participants who have been treated with oral anti hyperglycemia medications. Participants will receive 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes Mellitus (T2DM) for at least 1 year not treated with insulin
* Have been receiving at least two oral antihyperglycemic medications (OAMs) for at least 3 months prior to screening
* Have Hemoglobin A1c (HbA1c) of 7.0% to 11.0%, inclusive, according to central laboratory at screening
* Body mass index (BMI) ≤35.0 kilogram per square meter (kg/m^2)
* Inject insulin with a pre-filled insulin pen and perform Self-Monitored Blood Glucose (SMBG)
* Record keeping as required by this protocol
* Women of childbearing potential are not breastfeeding, have a negative pregnancy test at screening, do not plan to become pregnant during the study, have practiced reliable birth control during the study and 2 weeks following the last dose of investigational product

Exclusion Criteria:

* Have used insulin therapy (outside of pregnancy) anytime in the past 2 years, except for short term treatment of acute conditions
* Have been treated with rosiglitazone, pramlintide, glucagon-like peptide-1 (GLP-1) receptor agonist within 3 months prior to screening
* Are using or have used any of the following lipid-lowering medications: niacin preparations as a lipid-lowering medication and/or bile acid sequestrants within 90 days prior to screening
* Local OAM restrictions: have any restrictions for cardiac, renal, and hepatic diseases in the local product regulations
* Are taking, or have taken within 3 months before screening, prescription or over-the-counter medications to promote weight loss
* Have had any episodes of severe hypoglycemia, diabetic ketoacidosis, or hyperosmolar state/coma within 6 months prior to screening
* Have had 1 or more episodes of ketoacidosis or hyperosmolar state/coma in the past 6 months
* Have cardiac disease with functional status that is New York Heart Association Class III or IV
* Have a history of renal transplantation, or are currently receiving renal dialysis or have serum creatinine ≥2.0 milligram per deciliter (mg/dL) (177 micromole per liter [μmol/L]). Participants taking metformin should not exceed the creatinine level specified in the local label
* Have obvious clinical signs or symptoms of liver disease (excluding non-alcoholic fatty liver disease [NAFLD]), acute or any chronic hepatitis, non alcoholic steatohepatitis (NASH), or elevated liver enzyme measurements
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c
* Have active or untreated cancer, have been in remission from clinically significant cancer(other than basal cell or squamous cell skin cancer) for less than 5 years, or are at increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator
* Have known hypersensitivity or allergy to any of LY2605541 and insulin glargine or their excipients
* Have pre proliferative and proliferative retinopathy, maculopathy requiring treatment or not clinically stable in the last 6 months, or participants with active changes in subjective eye symptoms as determined by the investigator if an eye exam has not been performed in the last 6 months
* Are receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intranasal, intraocular, and inhaled preparations) or have received such therapy within the 8 weeks immediately preceding screening
* Have fasting triglycerides greater than 400 mg/dL (4.5 mmol/L) at screening as determined by the central laboratory
* Have an irregular sleep/wake cycle (for example, participants who sleep during the day and work during the night) in the investigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (31):
- Japan (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyazaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
- South Korea (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wŏnju
- Taiwan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sindian City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung County
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yongkang District
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhonghe

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Peglispro: Insulin Peglispro administered subcutaneously (SC) once daily for 26 weeks.
- Insulin Glargine: Insulin Glargine administered SC once daily for 26 weeks.
Period: Overall Study
Arm/Group | Insulin Peglispro | Insulin Glargine
Started | 192 | 196
Received at Least 1 Dose of Study Drug | 192 | 196
Completed | 182 | 186
Not Completed | 10 | 10
Not completed — Adverse Event | 2 | 3
Not completed — Protocol required discontinuation | 2 | 1
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Insulin Peglispro: Insulin Peglispro administered SC once daily for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Insulin Peglispro | Insulin Glargine | Total
Number analyzed (Participants) | 192 | 196 | 388
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 141 | 153 | 294
  >=65 years | 51 | 43 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 90 | 171
  Male | 111 | 106 | 217
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 192 | 196 | 388
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 103 | 102 | 205
  Taiwan | 40 | 42 | 82
  South Korea | 49 | 52 | 101
Baseline Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent of HbA1c] | 8.59 (1.09) | 8.48 (0.85) | 8.53 (0.97)
Fasting Serum Glucose (FSG) [Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)] | 165.11 (41.25) | 166.64 (36.81) | 165.88 (39.03)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Hemoglobin A1c (HbA1c)
Description: Hemoglobin A1c (HbA1c) is a test that measures a participant's average blood glucose level over the past 2 to 3 months. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis adjusting for treatment, stratification factors (region, sulfonylureas/meglitinide use, baseline Low-Density Lipoprotein [LDL-C], visit, treatment-by-visit interaction, and baseline HbA1c as fixed effects and participants as the random effect. P-value is from MMRM with terms for treatment, visit, treatment-by-visit interaction, stratification, and baseline HbA1C.
Time Frame: Baseline, Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable HbA1c data
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 179 | 184
percent of HbA1c | -1.61 (0.06) | -1.36 (0.06)
Statistical Analysis 1: Comparison: Insulin Peglispro vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — 0.4% is the margin of Non-inferiority; p = 0.005, Mixed Models Analysis; LS Mean Difference = -0.24, 95% CI 2-sided [-0.41 to -0.07]

2. Secondary Outcome: 30-Day Adjusted Rate of Total and Nocturnal Hypoglycemic Events
Description: Hypoglycemia Events (HE) occurs when blood glucose level ≤ 70 milligram per deciliter (mg/dL) (<3.9 micromoles per liter [mmol/L]). Nocturnal HE includes any total HE that occurred between bedtime and waking. Group mean rates of nocturnal hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models with treatment, baseline sulfonylurea/meglitinide use, baseline total hypoglycemia event rate, log (exposure/30 days) as the offset in the model. Group Mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline to Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable HE data.
Measure: Mean (Standard Error); unit: Number of events per participant per 30d
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 192 | 196
Number of events per participant per 30d
  Total HE | 1.28 (0.23) | 1.21 (0.23)
  Nocturnal HE | 0.19 (0.12) | 0.27 (0.18)

3. Secondary Outcome: Fasting Serum Glucose (FSG)
Description: LS means were calculated using MMRM analysis adjusting for baseline, treatment, stratification factor (region, HbA1c, LDL-C, and sulfonylurea [SU]/meglitinide use), visit, and treatment-by-visit interaction.
Time Frame: Weeks 0 and 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable FSG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 191 | 194
mg/dL
  Week 0 | 164.31 (2.78) | 166.61 (2.76)
  Week 26 | 103.85 (1.93) | 110.32 (1.90)

4. Secondary Outcome: Fasting Blood Glucose (FBG)
Description: LS Means were calculated using MMRM analysis adjusting for baseline, treatment, stratification factor (region, HbA1c, LDL-C, and SU/meglitinide use), visit and treatment-by-visit interaction.
Time Frame: Weeks 0 and 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable FBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 190 | 195
mg/dL
  Week 0 | 159.53 (2.51) | 161.19 (2.48)
  Week 26 | 108.39 (1.58) | 108.22 (1.55)

5. Secondary Outcome: Change From Baseline to Week 26 in Body Weight
Description: as for outcome 4
Time Frame: Baseline, Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 190 | 193
Kilogram (kg) | 1.06 (0.16) | 1.57 (0.16)

6. Secondary Outcome: 9-Point Self-Monitored Blood Glucose (SMBG)
Description: LS means were calculated using MMRM analysis adjusting for baseline, treatment, stratification factor (region, HbA1c, LDL-C, and SU/meglitinide use), visit and treatment-by-visit interaction. The 9-point SMBG are measured at: Pre-morning meal, 2 hours(hr) post morning meal, pre-midday meal, 2 hr post midday meal, pre-evening meal, 2 hr post pre-evening meal, bedtime, 0300 hr, and pre-morning meal next day, and should be performed on 2 non-consecutive days.
Time Frame: Week 0 and Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable SMBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 188 | 192
mg/dL
  Morning Pre-meal Wk0 | 160.19 (2.65) | 162.83 (2.62)
  Morning Pre-meal Wk26: number analyzed (Participants) | 176 | 183
  Morning Pre-meal Wk26 | 108.24 (1.68) | 108.71 (1.65)
  Morning Post-meal Wk0: number analyzed (Participants) | 185 | 189
  Morning Post-meal Wk0 | 237.19 (4.26) | 233.37 (4.21)
  Morning Post-meal Wk26: number analyzed (Participants) | 168 | 179
  Morning Post-meal Wk26 | 176.97 (3.31) | 176.93 (3.23)
  Mid-day Pre-meal Wk0: number analyzed (Participants) | 187 | 191
  Mid-day Pre-meal Wk0 | 169.24 (3.80) | 166.68 (3.76)
  Mid-day Pre-meal Wk26: number analyzed (Participants) | 171 | 181
  Mid-day Pre-meal Wk26 | 122.01 (2.56) | 122.85 (2.50)
  Mid-day Post-meal Wk0: number analyzed (Participants) | 186 | 188
  Mid-day Post-meal Wk0 | 224.22 (4.23) | 226.11 (4.21)
  Mid-day Post-meal Wk26: number analyzed (Participants) | 169 | 178
  Mid-day Post-meal Wk26 | 182.32 (3.26) | 183.88 (3.18)
  Evening Pre-meal Wk0: number analyzed (Participants) | 187 | 192
  Evening Pre-meal Wk0 | 176.49 (3.80) | 172.83 (3.75)
  Evening Pre-meal Wk26: number analyzed (Participants) | 171 | 182
  Evening Pre-meal Wk26 | 131.65 (3.08) | 135.55 (2.99)
  Evening Post-meal Wk0: number analyzed (Participants) | 185 | 189
  Evening Post-meal Wk0 | 219.45 (4.20) | 219.54 (4.16)
  Evening Post-meal Wk26: number analyzed (Participants) | 166 | 179
  Evening Post-meal Wk26 | 176.23 (3.37) | 182.80 (3.26)
  Bed Time Wk0: number analyzed (Participants) | 181 | 188
  Bed Time Wk0 | 198.64 (3.90) | 197.68 (3.83)
  Bed Time Wk26: number analyzed (Participants) | 167 | 177
  Bed Time Wk26 | 153.41 (2.95) | 161.44 (2.87)
  0300 Hours (Hrs) Wk0: number analyzed (Participants) | 176 | 179
  0300 Hours (Hrs) Wk0 | 158.82 (3.23) | 162.13 (3.20)
  0300 Hrs Wk26: number analyzed (Participants) | 156 | 167
  0300 Hrs Wk26 | 115.18 (2.34) | 114.77 (2.27)
  Pre-morning Meal Next Day Wk0: number analyzed (Participants) | 188 | 191
  Pre-morning Meal Next Day Wk0 | 156.28 (2.57) | 159.96 (2.55)
  Pre-morning Meal Next Day Wk26: number analyzed (Participants) | 176 | 181
  Pre-morning Meal Next Day Wk26 | 108.42 (1.73) | 105.18 (1.71)

7. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5%
Description: Percentage of participants with HbA1c ≤6.5% at Week 26 were made using a logistic regression model for endpoint used last observation carried forward (LOCF) method including treatment, baseline HbA1c value.
Time Frame: Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable HbA1c data.
Measure: Number; unit: Percentage of participants
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 191 | 194
Percentage of participants | 29.8 | 22.7

8. Secondary Outcome: Insulin Dose Per Kilogram (kg) of Body Weight
Description: LS means were calculated using MMRM analysis adjusting for baseline, treatment, stratification factor (region, HbA1c, LDL-C, and SU/meglitinide), visit, and treatment-by-visit interaction.
Time Frame: Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable insulin dose and body weight data.
Measure: Least Squares Mean (Standard Error); unit: units per kg
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 191 | 195
units per kg | 0.26 (0.01) | 0.26 (0.01)

9. Secondary Outcome: Percentage of Participants Achieving Steady-State of Basal Insulin Dose at 26 Weeks (Time to Steady State for Basal Insulin [Stable Maximum Dose])
Time Frame: Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable insulin dose data.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 192 | 196
percentage of participants | 96.9 | 97.2

10. Secondary Outcome: Concentration of Triglycerides, Total Cholesterol, Low-Density Lipoprotein (LDL-C), and High-Density Lipoprotein Cholesterol (HDL-C) at Week 26
Description: LS means were calculated using MMRM analysis adjusting for baseline, treatment, stratification factor (region, HbA1c, LDL-C, and SU/meglitinide use), visit, and treatment-by-visit interaction.
Time Frame: Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable laboratory data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 192 | 196
mg/dL
  Cholesterol Wk26: number analyzed (Participants) | 179 | 184
  Cholesterol Wk26 | 175.76 (1.65) | 177.90 (1.63)
  HDL Wk26: number analyzed (Participants) | 178 | 184
  HDL Wk26 | 51.64 (0.49) | 52.99 (0.48)
  Triglycerides Wk26: number analyzed (Participants) | 179 | 184
  Triglycerides Wk26 | 132.43 (4.71) | 122.83 (4.65)
  LDL Wk26: number analyzed (Participants) | 178 | 184
  LDL Wk26 | 97.95 (1.48) | 101.07 (1.46)

11. Secondary Outcome: Percentage of Participants With Detectable Anti-Insulin Peglispro Antibodies at Week 26
Description: For participants with detectable anti-insulin peglispro antibody level, the percentage of participants with positive cross-react with endogenous insulin was summarized.
Time Frame: Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable antibody data.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 192 | 196
percentage of participants | 24.6 | 32.5

12. Secondary Outcome: Change From Baseline of European Quality of Life-5 Dimensions - 3 Levels (EuroQoL-5D-3L ) Index Score and Visual Analog Scale (VAS) Health State Score at Week 26
Description: The EuroQoL-5D-3L questionnaire is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 3-level scale of 1 to 3 (no problem, some problems, and extreme problems). These combinations of attributes are converted into a weighted health-state Index Score according to the United States population-based algorithm. Scores ranged from -0.11 to 1.0 where a score of 1.0 indicates perfect health. Overall health state score was self-reported using a VAS marked on a scale of 0 to 100 (0 indicates worst imaginable health state and 100 indicates best imaginable health state. LS means were calculated using analysis of covariance (ANCOVA) for actual measures and changes from baseline at endpoint using LOCF method: adjusting for treatment, stratification factors (region, HbA1c and SU/meglitin.
Time Frame: Baseline, Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable EQ-5D data. Missing endpoints were imputed with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 184 | 192
units on a scale
  Change from Baseline to Endpoint EQ-5D-3L Score | 0.01 (0.01) | 0.00 (0.01)
  Change from Baseline VAS Health State Score | 2.29 (0.92) | 3.66 (0.90)

13. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ) Score
Description: The Insulin Treatment Satisfaction Questionnaire is a validated instrument containing 22 items that assessed treatment satisfaction for participants with diabetes on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, and Insulin Delivery Device. Data presented are the transformed score on a scale of 0-100, where a higher score indicate better treatment satisfaction. LS means was achieved using a MMRM model for post-baseline measures with stratification factors (country, HbA1c, and SU/meglitinide use) treatment, visit, treatment-by-visit as fixed effects. ITSQ was assessed at Week 4 (baseline) and Week 26.
Time Frame: Week 4 and 26
Population: All participants who were randomized and received at least 1 dose of study drug and have evaluable ITSQ data. Missing endpoints were imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 188 | 192
units on a scale
  ITSQ Wk4 | 74.13 (1.04) | 75.94 (1.03)
  ITSQ Wk26: number analyzed (Participants) | 179 | 184
  ITSQ Wk26 | 78.73 (1.06) | 78.29 (1.05)

14. Secondary Outcome: Change From Baseline to 26 Weeks in Adult Low Blood Sugar Survey (LBSS) Scores
Description: LBSS is a validated, participant-reported 33-item questionnaire with items rated on a 5-point Likert scale, where 0 = never and 5 - always. The LBSS measures behaviors to avoid hypoglycemia and its negative consequences (15 items) and worries about hypoglycemia and its negative consequences (18 items). Total score is the sum of all items (range 0 to 132). Higher total scores reflect greater fear of hypoglycemia. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country, treatment and metformin use as fixed effects and baseline score as a covariate. LBSS was assessed during screening visit (baseline) and again at Week 26.
Time Frame: Baseline, Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable LBSS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 184 | 192
units on a scale | 1.51 (0.69) | 1.62 (0.68)

15. Secondary Outcome: Intra-Participant Variability of the Fasting Blood Glucose (FBG)
Description: Intra-participant variability of Fasting Blood Glucose (FBG), which was measured by Self Monitored Blood Glucose (SMBG), was assessed by the standard deviation of the FBG measurement at the Week 26 visit. LS means were calculated using a MMRM with baseline fasting blood glucose measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Week 26
Population: All participants who were randomized and had at least 1 dose of study drug and had evaluable FBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 179 | 185
mg/dL | 14.97 (0.76) | 15.12 (0.75)

16. Secondary Outcome: Change From Baseline to 12 Weeks in Hemoglobin A1c (HbA1c)
Description: Hemoglobin A1c (HbA1c) is a test that measures a participant's average blood glucose level over the past 2 to 3 months.LS means were calculated using a MMRM with baseline HbA1C measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 191 | 194
percent of HbA1c | -1.43 (0.05) | -1.22 (0.05)

17. Secondary Outcome: Percent Hemoglobin A1c at Week 26
Description: HbA1c is a test that measures a participant's average blood glucose level over the past 2 to 3 months. LS means were calculated using a MMRM with baseline HbA1C measurement, stratification factors (country, HbA1c, LDL-C [< 100 mg/dL and ≥ 100 mg/dL], and SU/meglitinide use), treatment, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 191 | 194
percent of HbA1c | 6.92 (0.06) | 7.17 (0.06)

18. Secondary Outcome: Percentage of Participants With Total and Nocturnal Hypoglycemic Events (HE)
Description: Percentage of participants with hypoglycemic events (total or nocturnal) to Week 26 based on BG Threshold 70mg/dL.
Time Frame: Baseline to Week 26
Population: All participants who were randomized and received at least 1 dose of study drug and had evaluable HE data.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 192 | 196
percentage of participants
  Nocturnal Hypoglycemia BG 70mg/dL: number analyzed (Participants) | 51 | 58
  Nocturnal Hypoglycemia BG 70mg/dL | 26.6 | 29.6
  Total Hypoglycemia BG 70mg/dL: number analyzed (Participants) | 148 | 150
  Total Hypoglycemia BG 70mg/dL | 77.1 | 76.5

ADVERSE EVENTS:
Arm/Group | Insulin Peglispro | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 9/192 | 5/196
Other Adverse Events (participants affected / at risk) | 61/192 | 42/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=192) | Insulin Glargine (N=196)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Fracture treatment (Surgical and medical procedures) | 0 (0) | 1 (1)
Glaucoma surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Suprapubic prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=192) | Insulin Glargine (N=196)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (7) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 4 (5)
Gastroenteritis (Infections and infestations) | 4 (5) | 1 (2)
Nasopharyngitis (Infections and infestations) | 35 (46) | 29 (40)
Pharyngitis (Infections and infestations) | 8 (8) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 1 (1)
Weight increased (Investigations) | 6 (6) | 6 (6)
Headache (Nervous system disorders) | 6 (7) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No